CLINICAL TRIAL: NCT04868435
Title: Triggers for Post-Viral Parosmia After COVID-19 and Non-COVID-19 Infections
Brief Title: Triggers for Post-Viral Parosmia
Acronym: ParosmiaQ
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: AbScent (Unknown); University of London (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Jane Parker, Associate Professor, University of Reading
Other Study IDs: UoR SREC 29/2020
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Parosmia; Smell Disorder
Keywords: Parosmia; COVID; Trigger foods
MeSH Terms: conditions — Olfaction Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Many people lose their sense of smell after they have had a cold, flu or sinus infection. Recovery (if at all) generally starts with a "parosmia" phase which means every-day smells become distorted and over-poweringly objectionable, and this can lead to malnutrition and depression. We do not know much about how or why parosmia happens, but there are key foods common to those who suffer from parosmia which seem to trigger the distortion.

Parosmia and COVID-19 Loss of smell has recently been recognised as an official symptom of COVID-19, and we are starting to get reports of people who have recently had COVID-19 developing parosmia. The triggers seem to be similar to those of the common cold, flu or virus infections, but the journey between loss of smell and parosmia is different.

Hypotheses

1. Triggers of distortion will be the same for all parosmics.
2. There may be additional trigger foods in different cultures.

Questions

1. What are the trigger foods and beverages for parosmia?
2. Are there regional/cultural variations?
3. Does Covid-19 parosmia differ from "standard" post-viral parosmia?

The overall aim of the project is to understand the mechanisms involved in parosmia. The approach is to identify foods and everyday aromas associated with parosmia and to determine whether they are the same across different continents/cultures/ethnic backgrounds, and whether Covid-19 parosmia is any different to non-Covid-19 parosmia. The questionnaire will ask about Covid-19 status, ethnic background, smell loss and parosmia, and the changes that occurred between smell loss and parosmia. The participants will then answer questions on up to 15 everyday smells, some of which our preliminary evidence shows are common triggers, and others which are not. The questionnaire will be globally distributed, for example through current collaborations in the UK, US, Germany, Iran, China, Japan and Brazil. It will be completed by participants who are currently experiencing parosmia.

All participants will be asked to record any foods that they find distorted and provide a list of aromas which returned undistorted.

DETAILED DESCRIPTION:
The questionnaire will be sent out to those reporting early stages of parosmia as a result of post-viral infection, including post-COVID-19 infection. The questionnaire will record demographic data and ask about COVID-19 status, COVID-19 diagnosis and results of COVID-19 tests. It will ask about loss of smell, taste and chemesthesis (irritation from the heat of spices) and it will ask about the sequence of events leading to parosmia. Up to 15 everyday items will be rated for aroma description, intensity and valence. Participants will be asked to list other distorted foods, and also smells that returned undistorted. The questionnaire will be fully anonymous (unlinked anonymous) and voluntary. The questionnaire will be designed, distributed and data collected using the secure platform provided by Compusense.

ELIGIBILITY:
Inclusion Criteria:

* Individuals should be currently experiencing parosmia

Exclusion Criteria:

* Individuals below 18 years old will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be drawn from those currently suffering from parosmia only. Participants will initially be recruited from the AbScent membership which has a high proportion of UK and US members, but it will be rolled out internationally via ENT consultants.
Sampling Method: Non-Probability Sample
Enrollment: 943 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 20 minutes
  Outcomes from the questionnaire will be:
  List of major trigger foods for anosmia.
  Typical descriptions for smell distortions.
  Severity of parosmia.
  Patterns of anosmia/parosmia symptoms in post-viral infections including Covid-19.

CONTACTS AND LOCATIONS:
Overall Officials: Jane K Parker, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unlinked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- See also: Support and advice for those with smell disorders — http://abscent.org